CLINICAL TRIAL: NCT00475228
Title: Immediate Versus Delayed Insertion of the Levonorgestrel-Releasing Intrauterine Device Following Dilation and Evacuation: A Randomized Controlled Trial
Brief Title: 'Levonorgestrel IUD Insertion After D&E Procedure
Acronym: ILIAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Heather Hohmann, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pitt IRB PRO06040004
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Contraceptive Usage
Keywords: levonorgestrel IUD; IUD; dilation and evacuation; contraception
MeSH Terms: conditions — Contraception Behavior; Dilatation, Pathologic | interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Levonorgestrel IUD will be inserted immediately after completion of D&E
  Interventions: Drug: Levonorgestrel IUD
- Arm 2 (Active Comparator): Levonorgestrel IUD will be inserted at standard time post-procedure (3-6 weeks post D&E procedure)
  Interventions: Drug: Levonorgestrel IUD

INTERVENTIONS:
Drug: Levonorgestrel IUD — intrauterine insertion for arm 1 immediately after D&E procedure and for arm 2 at 3-6 weeks post-procedurem
  Other Names: Mirena

SUMMARY:
This study is a randomized controlled trial of insertion of the levonorgestrel-releasing intrauterine device (LNG-IUD) immediately following dilation & evacuation (D&E) compared to delayed insertion 3-6 weeks post-D&E. Eighty-eight women undergoing D&E between 15 0/7 and 23 6/7 weeks gestation will be enrolled at Magee-Womens Hospital, Pittsburgh, PA. The primary outcome is LNG-IUD usage six months following enrollment. We hypothesize that more women receiving immediate insertion will be using the LNG-IUD 6 months after the D&E procedure than women receiving delayed insertion. Secondary outcomes include the proportion receiving an IUD, continuation rate, complication rates, subject satisfaction, and quality of life. The utility of ultrasonography in predicting expulsion will also be examined. Anticipated problems include poor subject follow-up and coordinating the intra-operative study procedures.

DETAILED DESCRIPTION:
The D&E will be performed in the usual fashion. The uterus will be sounded to the fundus. Once the D&E is complete, the investigator or co-investigator will check the post-enrollment exclusion criteria to ensure that no events during the D&E made the subject ineligible. If the subject remains eligible, the randomization packet will be opened.

Immediately Post-D&E Procedure.

1. Group 1: IUD will be placed per study protocol. The strings will be trimmed to be flush with the cervix. Using transabdominal sonography, the distance from the serosal surface of the uterine fundus to the distal tip of the IUD will be measured.
2. Group 2: No additional procedures will be performed in the operating room.

Post-Operative Care. The subject will then be taken to the recovery room for routine post-operative care.

1. Group 1: A brief questionnaire will be administered. No additional procedures will be performed in the recovery room.
2. Group 2: A brief questionnaire will be administered. The subject will be asked to start her previously chosen method of contraception.
3. Subjects will be asked to call if any temperature exceeds 38°C (100.4°F). If a subject reports a fever (>38°C), an interim visit will be scheduled as described below.

Day 21-42. Post-D&E Visit at 1 month (PAV 1): will be scheduled on a weekday between 8:30 am and 4:30 pm at the time most convenient for the subject. For Group 1, the visit may be on any day from day 21-42. For Group 2, the visit will be scheduled with the goal of inserting the LNG-IUD during the first 7 days of the menstrual cycle.

Subjects will complete a questionnaire about symptoms since the D&E, including pain and bleeding and subjects' history will be collected. Subjects also will complete a set of visual-analog scales about pain, bleeding, and quality of life. All subjects will have a bimanual exam to assess uterine size, cervical motion and adnexal tenderness. Women in Group 1 will have a speculum exam to measure and, if necessary, trim the IUD strings. The length of the segment trimmed will be measured and recorded. If cervicitis or vaginitis is suspected, further evaluation will be performed with diagnosis and treatment by CDC guidelines as indicated. Women in group 2 will have their IUD placed.

Day 56-70: Post-D&E Visit at 2 months (PAV 2): may be scheduled any time within days 56-70 but must be at least 21 days after PAV1. Subjects will complete a questionnaire and visual-analog scales about symptoms since the D&E, including pain, bleeding, and quality of life and subjects' history will be obtained. Bimanual Examination will be performed to assess uterine size, cervical motion and adnexal tenderness. A speculum exam will be done to measure the strings and trim, if necessary. The IUD-Fundal Distance will be assessed by endovaginal sonography.

Day 160-200: Telephone Interview at 6 month (TI 6). A questionnaire will be administered over the phone. Three attempts will be made to contact the subject by telephone. A certified letter with the questionnaire and a postage-paid envelope will be sent if the subject is not contacted.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age from 15 weeks 0 days to 23 weeks 6 days at enrollment (time of D&E), confirmed by ultrasound
2. Has already consented to a D&E
3. Desires to use the LNG-IUD (Mirena) for contraception for 12 months or more
4. Willing and able to sign an informed consent
5. Willing to comply with the study protocol
6. Age greater than or equal to 18 years
7. Primary residency in Allegheny, Beaver, Washington, Westmoreland, Butler, Armstrong, Indiana, Fayette, Greene, or Lawrence counties of Pennsylvania

Exclusion Criteria:

1. Allergy to either polyethylene or levonorgestrel
2. Urgent need for termination of pregnancy (active bleeding or infection)
3. Exposure to or treatment for gonorrhea or Chlamydia within the past 90 days
4. Diagnosis of pelvic inflammatory disease within the past year
5. Presence of one or more leiomyomata greater than 3 centimeters in diameter
6. Uterine anomaly (other than a repaired septate uterus)
7. Current participation in any other intervention trial

Post-Enrollment Pre-Randomization Exclusion criteria (to be assessed at the completion of the D&E. These criteria will be used to define a group not eligible for immediate insertion. Since these complications contraindicate immediate insertion, the issue of whether immediate and delayed insertion is preferable is no longer in question.)

1. Uterine perforation
2. Hemorrhage as defined by one of the following: (1) need for transfusion; (2) estimated blood loss greater than 500 cc; (3) intrauterine placement of a Foley catheter; or (4) the use of 3 or more doses of uterotonic medications
3. Evidence of infection at the time of the D&E, including fever (temperature ≥ 38°C) or pus at the cervical os
4. Subject no longer desires a LNG-IUD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2007-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hohmann, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Center for Family Planning Research, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Women undergoing D&E at 15 to 23 weeks of gestation were approached for enrollment. After completion of the D&E, women who consented were enrolled as long as there no contraindications to immediate IUD insertion. 88 out of the 93 subjects were randomized to either Arm I (immediate) or Arm 2 (delayed, 3 to 6 weeks later LNG-IUD insertion).
Groups:
- Arm I: Immediate LNG-IUD Insertion Group: Levonorgestrel IUD will be inserted immediately after completion of D&E
  Levonorgestrel IUD: intrauterine insertion for arm 1 immediately after D&E procedure and for arm 2 at 3-6 weeks post-procedurem
- Arm 2: Delayed (3-6 Weeks) LNG-IUD Insertion Group: Levonorgestrel IUD will be inserted at standard time post-procedure (3-6 weeks post D&E procedure)
  Levonorgestrel IUD: intrauterine insertion for arm 1 immediately after D&E procedure and for arm 2 at 3-6 weeks post-procedurem
Period: Overall Study
Arm/Group | Arm I: Immediate LNG-IUD Insertion Group | Arm 2: Delayed (3-6 Weeks) LNG-IUD Insertion Group
Started | 44 | 44
Completed | 27 | 27
Not Completed | 17 | 17
Not completed — Lost to Follow-up | 17 | 17

BASELINE CHARACTERISTICS:
Population: After completion of the D&E, 88 of the 93 women who consented were randomized 1:1 to Arm 1 and Arm 2.
Groups:
- Arm I: Immediate LNG-IUD Insertion Group: Subjects randomized to Arm I had the Levonorgestrel IUD placed using ultrasound guidance immediately after completion of D& E
- Arm 2: Delayed LNG-IUD Insertion Group: Subjects randomized to Arm 2 had the Levonorgestrel IUD placed at 3 to 6 weeks post-procedure as per standard of care practice.
- Total: Total of all reporting groups
Arm/Group | Arm I: Immediate LNG-IUD Insertion Group | Arm 2: Delayed LNG-IUD Insertion Group | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Customized [Number; unit: participants]
  at least 18 years of age | 44 | 44 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is LNG-IUD Usage Six Months Following Enrollment.
Description: To assess the six-month usage rate of the LNG-IUD when placed immediately after D&E compared to 3-6 weeks later, as measured by the proportion of women with a LNG-IUD in place at six months after the D&E.
  We hypothesize that more women receiving immediate insertion will be using the LNG-IUD 6 months after the D&E procedure than women receiving delayed insertion.
Time Frame: 6 months
Population: Attempts to contact all participants (Arm 1: 44 women and Arm 2: 44 women) by phone 6 months post D&E were made. For Arm 1, 27 out of 44 women could be reached. For Arm 2; 27 out of the 44 were reached (19 women who returned and had the LNG-IUD placed 3-6 weeks post D&E and 8 women who did not return for the LNG-IUD placement 3-6 post D&E).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Immediate LNG-IUD Insertion Group | Arm 2: Delayed (3-6 Weeks) LNG-IUD Insertion Group
Number analyzed (Participants) | 27 | 27
percentage of participants | 85.2 [66.3 to 95.8] | 62.9 [42.4 to 80.6]
Statistical Analysis 1: Comparison: Arm I: Immediate LNG-IUD Insertion Group vs Arm 2: Delayed (3-6 Weeks) LNG-IUD Insertion Group; Test type: Superiority or Other; p = 0.05, Chi-squared

2. Secondary Outcome: To Examine the Number of Women Receiving the LNG-IUD in Each Group
Description: The difference between the overall number of women who had the LNG-IUD inserted immediately post D&E successfully (Arm 1) was compared to the overall number of women who had the LNG-IUD inserted 3 -6 weeks post D&E (standard or routine) (Arm 2).
Time Frame: 2 Months
Population: In Arm 1, all 44 participants were inserted with an LNG-IUD immediately post D& E successfully. In Arm 2; only 20 of the 44 participants returned and had the LNG-IUD inserted successfully 3 to 6 weeks post D&E.
Measure: Number; unit: Completed LNG-IUD Insertions
Units Other Than Participants: Completed LNG-IUD Insertions
Groups:
- Arm 2: Delayed (3-6 Weeks) LNG-IUD Insertion Group: Levonorgestrel IUD was inserted at standard time post-procedure (3-6 weeks post D&E procedure) in 20 participants. The remaining 24 women did not return 3-6 weeks after the D&E.
  Levonorgestrel IUD: intrauterine insertion for arm 1 immediately after D&E procedure and for arm 2 at 3-6 weeks post-procedurem
- Arm I: Immediate LNG-IUD Insertion Group: Levonorgestrel IUD was inserted immediately after completion of D&E in all 44 participants
  Levonorgestrel IUD: intrauterine insertion for arm 1 immediately after D&E procedure and for arm 2 at 3-6 weeks post-procedurem
Arm/Group | Arm 2: Delayed (3-6 Weeks) LNG-IUD Insertion Group | Arm I: Immediate LNG-IUD Insertion Group
Number analyzed (Participants) | 44 | 44
Number analyzed (Completed LNG-IUD Insertions) | 20 | 44
Completed LNG-IUD Insertions | 20 | 44

3. Secondary Outcome: To Compare Expulsion Rates Between Immediate Insertion and Delayed Insertion
Description: Compared the expulsion rate of the LNG-IUD in the participants who received the LNG-IUD in the immediate and delayed insertion group
Time Frame: 6 months
Population: 3 of the 44 participants who had the LNG-IUD placed in Arm 1 underwent an IUD expulsion. 1 of the 20 participants who had the LNG-IUD placed in Arm 2 underwent an IUD expulsion.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I: Immediate LNG-IUD Insertion Group | Arm 2: Delayed LNG-IUD Insertion Group
Number analyzed (Participants) | 44 | 20
percentage of participants | 6.8 | 5.0

ADVERSE EVENTS:
Time Frame: Adverse data related to expulsion collected from the time of the IUD insertion and up to 6 months.
Arm/Group | Arm I | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No